CLINICAL TRIAL: NCT05567094
Title: The Effect of Perioperative DEXamethasone on Postoperative Complications After PANcreaticoduodenectomy
Acronym: PANDEX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, BAIYONG SHEN, Professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PANDEX-1
Record Dates: First submitted 2022-09-30; First posted 2022-10-05 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Pancreaticoduodenectomy
Keywords: Pancreaticoduodenectomy; Dexamethasone; Postoperative complications; Double-blind; Pragmatic; Superiority trial
MeSH Terms: conditions — Postoperative Complications | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive 0.2 mg/kg dexamethasone or saline placebo, administered as an intravenous bolus within 5 minutes after induction of anesthesia.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patients, surgeons, anesthetists, data collectors, and outcome assessors are all blinded. Only the data manager and the specific study coordinator are unblinded to the group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone (Experimental): Patients will receive 0.2 mg/kg dexamethasone, administered as an intravenous bolus within 5 minutes after induction of anesthesia
  Interventions: Drug: Dexamethasone
- Saline placebo (Placebo Comparator): Patients will receive 2ml saline placebo, administered as an intravenous bolus within 5 minutes after induction of anesthesia
  Interventions: Drug: Saline placebo

INTERVENTIONS:
Drug: Dexamethasone — Patients will receive 0.2 mg/kg dexamethasone, administered as an intravenous bolus within 5 minutes after induction of anesthesia
  Arms: Dexamethasone
Drug: Saline placebo — Patients will receive 2ml saline placebo, administered as an intravenous bolus within 5 minutes after induction of anesthesia
  Arms: Saline placebo

SUMMARY:
The primary objective of this clinical trial is evaluate the effect of dexamethasone on postoperative complications after pancreaticoduodenectomy.

DETAILED DESCRIPTION:
This is a multicentric, prospective, randomized, double-blind, pragmatic, placebo-control study. Patients who are going to receive elective pancreaticoduodenectomy will be randomized to receive 0.2 mg/kg dexamethasone or saline placebo, administered as an intravenous bolus within 5 minutes after induction of anesthesia. The primary outcome is the Comprehensive Complication Index (CCI) score within 30 days after the operation, which will be compared between these two groups .

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients ≥18 years of age;
2. An indication for elective PD surgery;
3. Patients understand the nature of this trial and are willing to comply;
4. Patients are able to provide written informed consent;

Exclusion Criteria:

1. Current or recent (within preceding 1 month) systemic use of glucocorticoids;
2. Distant metastases including peritoneal carcinomatosis, liver metastases, distant lymph node metastases, and involvement of other organs;
3. Patients may undergo left, central, or total pancreatectomy other than PD;
4. Palliative surgery；
5. Patients with high operative risk, as defined by the American Society of Anesthesiologists (ASA), with a score ≥ 4;
6. Synchronous malignancy in other organs or second cancer requiring resection during the same procedure;
7. Pregnant and lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2022-10-08 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
The Comprehensive Complication Index (CCI) | Within 30 days after the operation
  The Comprehensive Complication Index (CCI) score within 30 days after the operation.
  The CCI takes into account all cumulative complications and receives values between 0 and 100. The weight of complication (wC) of the CCI is based on the established Clavien-Dindo classification.

SECONDARY OUTCOMES:
The incidence of major complications (Clavien-Dindo≥3) | 30 days
The incidence of postoperative pancreatic fistula (ISGPS classification) | 30 days
The incidence of postpancreatectomy acute pancreatitis (ISGPS classification) | 30 days
The incidence of infection (including wound infection and intra-abdominal abscess) | 30 days
Postoperative length of stay | 1 day of discharge
The incidence of relaparotomy | 30 days
Mortality | 30 days
Mortality | 60 days

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen H, Wang C, Shen Z, Wang W, Weng Y, Ying X, Deng X, Shen B. Postpancreatectomy Acute Pancreatitis After Pancreaticoduodenectomy: A Distinct Clinical Entity. Ann Surg. 2023 Aug 1;278(2):e278-e283. doi: 10.1097/SLA.0000000000005605. Epub 2022 Jul 18. PMID 35848748
- [Background] DREAMS Trial Collaborators and West Midlands Research Collaborative. Dexamethasone versus standard treatment for postoperative nausea and vomiting in gastrointestinal surgery: randomised controlled trial (DREAMS Trial). BMJ. 2017 Apr 18;357:j1455. doi: 10.1136/bmj.j1455. PMID 28420629
- [Background] Corcoran TB, Myles PS, Forbes AB, Cheng AC, Bach LA, O'Loughlin E, Leslie K, Chan MTV, Story D, Short TG, Martin C, Coutts P, Ho KM; PADDI Investigators; Australian and New Zealand College of Anaesthetists Clinical Trials Network; Australasian Society for Infectious Diseases Clinical Research Network. Dexamethasone and Surgical-Site Infection. N Engl J Med. 2021 May 6;384(18):1731-1741. doi: 10.1056/NEJMoa2028982. PMID 33951362
- [Background] Laaninen M, Sand J, Nordback I, Vasama K, Laukkarinen J. Perioperative Hydrocortisone Reduces Major Complications After Pancreaticoduodenectomy: A Randomized Controlled Trial. Ann Surg. 2016 Nov;264(5):696-702. doi: 10.1097/SLA.0000000000001883. PMID 27429037
- [Background] Asehnoune K, Le Moal C, Lebuffe G, Le Penndu M, Josse NC, Boisson M, Lescot T, Faucher M, Jaber S, Godet T, Leone M, Motamed C, David JS, Cinotti R, El Amine Y, Liutkus D, Garot M, Marc A, Le Corre A, Thomasseau A, Jobert A, Flet L, Feuillet F, Pere M, Futier E, Roquilly A; PACMAN study group. Effect of dexamethasone on complications or all cause mortality after major non-cardiac surgery: multicentre, double blind, randomised controlled trial. BMJ. 2021 Jun 2;373:n1162. doi: 10.1136/bmj.n1162. PMID 34078591
- [Derived] Chen H, Wang Y, Wang C, Lu X, Li Y, Sun B, Jiang K, Qiu Y, Chen R, Cao L, Chen S, Luo Y, Shen B. The effect of perioperative of dexamethasone on postoperative complications after pancreaticoduodenectomy (PANDEX): a study protocol for a pragmatic multicenter randomized controlled trial. Trials. 2023 Sep 2;24(1):569. doi: 10.1186/s13063-023-07571-y. PMID 37660052